CLINICAL TRIAL: NCT06633120
Title: In Vitro Maturation of Human Eggs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado Center for Reproductive Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20141020
Record Dates: First submitted 2024-09-25; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Healthy; PCOS; PCOS (Polycystic Ovary Syndrome); Ovarian Reserve; Infertility; Infertility Female; Infertility of Tubal Origin; Infertility Poly Cystic Ovary; AMH; In Vitro Maturation; IVM; IVF
Keywords: IVM; Infertility; PCOS; IVF
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility; Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Biphasic IVM Treatment (Experimental): Biphasic IVM of oocytes
  Interventions: Other: IVM

INTERVENTIONS:
Other: IVM — Immature oocytes will be retrieved from small ovarian follicles and matured overnight in the laboratory prior to undergoing fertilization and embryo culture.

SUMMARY:
CCRM Fertility, a global pioneer in fertility treatment, research and science, is seeking participants for a new study on in vitro maturation (IVM). IVM requires less hormones to stimulate the ovaries than IVF, making it more affordable than IVF with fewer side effects. Participants that qualify for the study will receive a free cycle of IVM treatment at CCRM Fertility and including a new patient consultation, fertility testing, preimplantation genetic testing for aneuploidies (PGT-A), anesthesia and some medication

DETAILED DESCRIPTION:
Patients will undergo a complete IVF workup to qualify for study. Once passing their baseline appointment patients will undergo a three day low dose stimulation followed by egg retrieval 18-22 hours post last medication dosage. Immature oocytes will be retrieved from the ovaries via ultrasound guided TV aspiration and matured overnight in the laboratory. Mature oocytes will be fertilized via ICSI the following day and cultured to the blastocyst stage. Biopsy of the first 14 blastocysts are included with this package, patients have the option biopsy additional embryos if available. Biopsies will be sent for PGTA testing. This study also includes preparation for and the first frozen embryo transfer. Some FET medication is included as well as testing through the first pregnancy test.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women diagnosed with PCOS or polycystic ovaries, or infertile women with good ovarian reserve
* Antral follicle count (AFC) greater than 24
* AMH greater than 3.5 ng/ml
* Body Mass Index less than 35
* Accept to have embryos biopsied for PGT
* Intend to perform embryo transfer within 4 months after completing the IVM cycle
* Paternal (or donor) age <45, ejaculated sperm collection only (partner frozen and donor sperm acceptable), sperm morphology (strict criteria) >1%, motility > 20% and sperm count > 10 million per ml (so samples can be prepared through standard procedure)

Exclusion Criteria:

* More than 2 failed IVF cycles

Max Age: 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Oocyte maturation | 27 hours
  Maturation rate of retrieved oocytes
Embryo fertilization and development | 7 days
  Number of embryos that fertilize and develop after ICSI. Blastocysts will be biopsied and frozen on days 5, 6, and 7 of development
Pregnancy | 6 months
  Pregnancy following embryo transfer. HCG levels and ultrasound confirming IUP and heartrate.

SECONDARY OUTCOMES:
Live Birth | 12 months
  Birth information (sex of infant, status, weight, and any complications) will be collected via patient contact when possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado Center for Reproductive Medicine, Lone Tree, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared through publication in scientific journals.